CLINICAL TRIAL: NCT01766310
Title: Effect of Folic Acid Supplementation on Plasma Homocysteine Level in Obese Children: a Randomized Double Blinded Placebo Controlled Trial
Brief Title: Effect of Folic Acid Supplementation on Plasma Homocysteine Level in Obese Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pavinee Intakorn, Queen Sirikit National Institute of Child Health, Queen Sirikit National Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Folic-01
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Hyperhomocysteinemia; Obesity
Keywords: Folic acid; Folate; Homocysteine; Obese; Children
MeSH Terms: conditions — Hyperhomocysteinemia; Obesity | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo tablet in the same appearance and taste with folic acid orally once a day for 8 weeks of the study
  Interventions: Drug: placebo
- folic acid (Experimental): Folic acid tablet 5mg per day orally (5mg/tablet) once a day for 8 weeks of the study
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Folic Acid — yellow tablet contained 5mg of folic acid, manufactured from the Government Pharmaceutical Organization, Ministry of Public Health, Thailand
  Arms: folic acid
Drug: placebo — sugar tablet manufactured to mimic folic acid tablet
  Arms: placebo

SUMMARY:
The purpose of the present study was to determine whether folic acid supplementation could reduce plasma homocysteine in obese children and to determine the association between dietary folate, serum folate and homocysteine level through the randomized double blinded placebo controlled trial.

DETAILED DESCRIPTION:
Atherosclerosis is common & remains a significant clinical problem because of leading to myocardial infarction, stroke and cardiovascular death. Many studies founded hyperhomocysteinemia is an independent risk factor for those cardiovascular diseases which take responsible for about 10% of total cardiovascular disease risk. Reduction of elevated plasma homocysteine may prevent up to 25% of cardiovascular events. One of modifiable cause of hyperhomocysteinemia is prevention of vitamin deficiency, especially folate deficiency.

Obese Thai children are probable risk for folate deficiency due to low dietary folate intake and low serum folate level from unbalanced diet (low vegetables intake & high fat diet) and high prevalence of thalassemia. Moreover obese children are also at risk of atherosclerosis. However, no data have been reported about effect of folic acid supplementation on homocysteine level in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 9-18 years
* Diagnosed obesity (BMI more than median plus two of standard deviation for age and sex according to WHO reference 2007)

Exclusion Criteria:

* Secondary obesity
* Thalassemia disease
* Renal and hepatic dysfunction
* Drugs: anticonvulsant, estrogen, thiazides, metformin, cholestyramine, methotrexate, fibrates, nicotinic acid
* Previous vitamin supplementation 1 month before study

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orawan Iamopas, MD., Principal Investigator — Queen Sirikit National Institute of Child Health
Locations (2):
- Thailand (2):
  - Department of Pediatrics, Queen Sirikit National Institute of Child Health, Bangkok, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok, Bangkok

REFERENCES:
- [Background] Solini A, Santini E, Ferrannini E. Effect of short-term folic acid supplementation on insulin sensitivity and inflammatory markers in overweight subjects. Int J Obes (Lond). 2006 Aug;30(8):1197-202. doi: 10.1038/sj.ijo.0803265. Epub 2006 Feb 21. PMID 16491109
- [Background] Papandreou D, Malindretos P, Arvanitidou M, Makedou A, Rousso I. Oral supplementation of folic acid for two months reduces total serum homocysteine levels in hyperhomocysteinemic Greek children. Hippokratia. 2010 Apr;14(2):105-8. PMID 20596265
- [Background] Papandreou D, Malindretos P, Arvanitidou M, Makedou A, Rousso I. Homocysteine lowering with folic acid supplements in children: effects on blood pressure. Int J Food Sci Nutr. 2010 Feb;61(1):11-7. doi: 10.3109/09637480903286371. PMID 19939196
- [Background] Pena AS, Wiltshire E, Gent R, Hirte C, Couper J. Folic acid improves endothelial function in children and adolescents with type 1 diabetes. J Pediatr. 2004 Apr;144(4):500-4. doi: 10.1016/j.jpeds.2003.12.049. PMID 15069400
- [Background] Gargari BP, Aghamohammadi V, Aliasgharzadeh A. Effect of folic acid supplementation on biochemical indices in overweight and obese men with type 2 diabetes. Diabetes Res Clin Pract. 2011 Oct;94(1):33-8. doi: 10.1016/j.diabres.2011.07.003. Epub 2011 Jul 28. PMID 21802161
- [Derived] Iamopas O, Ratanachu-ek S, Chomtho S. Effect of folic acid supplementation on plasma homocysteine in obese children: a randomized, double-blind, placebo-controlled trial. J Med Assoc Thai. 2014 Jun;97 Suppl 6:S195-204. PMID 25391194

RESULTS

PARTICIPANT FLOW:
Groups:
- Folic Acid: Folic acid tablet 5mg per day orally (5mg/tablet) once a day for 8 weeks of the study
  Folic Acid
Period: Overall Study
Arm/Group | Placebo | Folic Acid
Started | 24 | 26
Completed | 23 | 23
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: mean and SD
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Folic Acid | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.73 (1.64) | 11.08 (1.57) | 10.90 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes of Homocysteine Level
Description: Mean difference of changes of homocysteine level between 2 treatment groups
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo | Folic Acid
Number analyzed (Participants) | 23 | 23
µmol/L | -0.68 (1.25) | -1.35 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Folic Acid; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Net) = 0.68, 95% CI 2-sided [-0.09 to 1.44], Standard Deviation 1.3

2. Secondary Outcome: Serum Folate Level
Description: correlation between serum folate and plasma homocysteine level
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Serum Vitamin B12 Level
Description: correlation between serum vitamin B12 and plasma homocysteine level
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Prevalence of Hyperhomocysteinemia
Description: prevalence of hyperhomocysteinemia in Thai obese children
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Placebo | Folic Acid
Number analyzed (Participants) | 24 | 26
participants | 3 | 2

ADVERSE EVENTS:
Arm/Group | Placebo | Folic Acid
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No